CLINICAL TRIAL: NCT01573156
Title: Vascular Targeted Photodynamic Therapy With WST11 for T1a Renal Tumours. PHASE IIa Histological Follow up Trial
Brief Title: Vascular Targeted Photodynamic Therapy T1a Renal Tumours
Acronym: KCM201
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Concerns about post VTP MRI results being conclusive
Sponsor: University of Oxford (Other)
Collaborators: Steba Biotech S.A. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN1102 KCM201; 2011-003311-27 (EudraCT Number)
Record Dates: First submitted 2012-03-22; First posted 2012-04-06 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Renal Cancer
Keywords: renal cancer; photodynamic therapy; wst 11
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VTP treatment to small renal mass (Experimental)
  Interventions: Drug: Light activated WST11

INTERVENTIONS:
Drug: Light activated WST11 — WST11-mediated VTP will consist of the combination of a single IV administration of WST11 at doses of 2 mg/kg, or 4mg/kg using 753 nm laser light at a fixed power (150 mW/cm) and energy (200 J/cm) delivered through percutaneous optical fibres. The fibres are introduced into transparent needles that are positioned in the areas of interest under CT image guidance. After a minimum of 3 patients at each drug dosage (2 & 4 mg/kg) has been treated with a light energy of 200 J/cm, the general and local safety will be assessed. The safety results of the first 3 patients treated in each drug dose/number of fibres combination will be reviewed by the investigators prior to escalation to a higher drug dose/number of fibres combination.
  Other Names: Tookad Soluble

SUMMARY:
Vascular Targeted Photodynamic therapy (VTP) with the Vascular Occluding Agent (VOA) WST11, may offer an alternative, providing tumour destruction via a minimally invasive approach. In this investigation, the investigators plan to use the WST11 VTP procedure to treat a predetermined small renal tumour targets. Patients will be given a general anaesthetic, to ensure immobility, and prevent discomfort during treatment sessions. Treated patients will then undergo surgical resection of their tumours, and the accuracy and reliability of tissue death with VTP will be assessed histologically. The aim of this proof of concept study is to demonstrate whether this modality has potential for a clinical role in the treatment of oncological kidney disease, either as an alternative to surgery, or where surgery is not feasible.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or post-menopausal female, aged 60 years or above.
* Lesions suspicious for renal cell carcinoma on triple phase CT that are < 4cm in maximum diameter and suitable for surgical resection
* Participant must be in sufficiently good health to be suitable for general anaesthesia for both VTP treatment and subsequent surgical resection of tumour
* Subjects must have ≥ 1 evaluable tumours which can be visualized on diagnostic ultrasound. If more than one tumour exists, an index tumour will be nominated and treated (uncommon)
* Previous chemotherapy and / or biological therapy for cancer are permitted, but the subject should have recovered fully from the effects of these and any prior surgery (minimum of 28 days).
* Patients should not have received radiotherapy to the target area within the preceding 12 months.
* Subject has clinically acceptable haematological, electrolyte and hepatic function as demonstrated by serum laboratory values within 14 days prior of VTP treatment:
* Absolute neutrophil count (ANC) ≥ 1500mm-3
* Platelet count ≥ 100,000mm-3
* Haemoglobin ≥ 10gdl-1
* Prothrombin time (PT) ≤ 1.5 * Upper Limit of Normal (ULN)
* Activated partial thromboplastin time (APPT) ≤ 1.5 * ULN
* Total bilirubin < 2.5 * ULN
* Aspartate aminotransferase (AST) < 3 * ULN
* Alkaline phosphatase (ALP) < 2 * ULN; unless arising from bone
* Participants has a clinically acceptable ECG
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Non menopausal women
* Significant hepatic impairment.
* Significant renal impairment as to mean surgical resection is unsuitable
* Clinical or radiological evidence of metastatic disease
* Subjects with tumours lying adjacent to vital structures such that VTP treatment would risk damage to these structures
* Subjects currently taking immunosuppressive medication
* Patients whose medical conditions need the following medication which have potential photosensitizing effects (tetracyclines, sulphonamides, phenothiazines, sulfonylurea hypoglycaemic agents, thiazide diuretics, griseofulvin and amiodarone (see appendix G)) if these treatments cannot be stopped or replaced by other treatments without photosensitizing properties
* Patients who have an absolute need for anticoagulant drugs or antiplatelet drugs (e.g., warfarin, aspirin), which cannot be withdrawn during the 10 days prior to the VTP procedure.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Participants involved in the treatment phase of a clinical trial (observational or follow-up studies will be allowed)
* An American Society of Anaesthesiologists (ASA) score of ≥ 3
* A World Health Organization (WHO) performance status of ≥2

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Volume of tumour necrosis on final histology expressed as a percentage of pre-treatment tumour volume | 2-4 weeks post VTP therapy

SECONDARY OUTCOMES:
Radiological evidence of tissue destruction at day 12 (technical success) based on the volume of tumour ablation on day 12 MRI imaging expressed as a percentage of pre-treatment tumour volume | 12 days post VTP therapy
Adverse events according to Common Toxicity Criteria (CTCAE) | Up to 12 months post VTP

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sullivan, MD FRCS Urol, Principal Investigator — Churchill Hospital, Oxford, UK
Locations (1):
- Churchill Hospital, Oxford, United Kingdom